CLINICAL TRIAL: NCT01615406
Title: A Phase 1 Pilot Comparison Study of 99mTc-MIP-1404 Single Photon Emission Computed Tomography (SPECT)/CT Imaging to Histology in Men With Prostate Cancer
Brief Title: A Phase 1 Pilot Study of 99mTc-MIP-1404 SPECT/CT Imaging to Histology in Men With Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Molecular Insight Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MIP-1404-P105
Record Dates: First submitted 2012-06-04; First posted 2012-06-08 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — technetium 99m 1-(1-(2-(bis(carboxymethyl)amino)-2-oxoethyl)-1H-imidazol-2-yl)-2-((1-(2-(bis(carboxymethyl)amino)-2-oxoethyl)-1H-imidazol-2-yl)methyl)-9,14-dioxo-2,8,13,15-tetraazaoctadecane-7,12,16,18-tetracarboxylic acid)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Drug: 99mTc-MIP-1404 (Experimental): 20 ±3 mCi intravenous (IV) injection of 99mTc MIP 1404
  Interventions: Drug: 99mTc MIP 1404

INTERVENTIONS:
Drug: 99mTc MIP 1404 — A single dose of 20 ±3 mCi intravenous (IV) injection of 99mTc MIP 1404

SUMMARY:
This is a single arm, open label study of up to 24 prostate cancer patients scheduled for prostatectomy and/or pelvic lymph node dissection. Patients receive a single IV dose of 99mTc-MIP-1404 (study drug) followed by SPECT/CT scan 3-6 hours after injection. As standard of care, patients will undergo prostatectomy and/or pelvic lymph node dissection (PLND) within two weeks of study drug dosing. 99mTc-MIP-1404 image data will be evaluated for visible uptake and compared with histopathology.

ELIGIBILITY:
Inclusion Criteria:

* Male aged 21 years or older.
* Ability to provide signed informed consent and willingness to comply with protocol requirements.
* Past biopsy indicating the presence of adenocarcinoma of the prostate gland.
* Participant is deemed to have tissue suspicious of prostate cancer involvement that is amenable to biopsy/resection.
* Have had, or will undergo diagnostic CT or MRI imaging prior to surgery.
* Participants must agree to use an acceptable form of birth control throughout the study period. Participants must use condoms for a period of seven days after study drug administration, if engaged in sexual activity.

Exclusion Criteria:

* Participants for whom participating would significantly delay the scheduled standard of care therapy.
* Participants administered a radioisotope within 5 physical half lives prior to study enrollment.
* Participants with any medical condition or other circumstances that, in the opinion of the investigator, would significantly decrease obtaining reliable data, achieving study objectives or completing the study.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-04; Primary Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Tissue distribution of 99mTc-MIP-1404 SPECT/CT imaging in tumor and non-tumorous regions of the prostate | Within 3-6 hours of dosing SPECT/CT images will be taken
  Tissue distribution of 99mTc-MIP-1404 SPECT/CT imaging in tumor and non-tumorous regions of the prostate (as determined by histopathology) in patients undergoing standard of care prostatectomy

SECONDARY OUTCOMES:
Safety of 99mTc-MIP-1404 will be assessed by measuring Vital Signs (blood pressure and heart rate)Pre-Dose and Post-Dose as well as between 3-6 hours post-dose | Vital signs measurements will be taken, an expected average of 30 minutes before and after study drug injection and between 3-6 hours after study drug injection
  Summary tables will present change from pre-dose to post-dose vital signs measurements.
Tissue distribution of 99mTc-MIP-1404 SPECT/CT imaging in tumor and non-tumorous regions of pelvic lymph node | Within 3-6 hours of dosing SPECT/CT images will be taken
  To obtain exploratory tissue distribution of 99mTc-MIP-1404 SPECT/CT imaging in tumor and non-tumorous regions of pelvic lymph node
Intensity of 99mTc-MIP-1404 uptake with respect to PSMA expression | PSMA expression analysis will be conducted upon completion of enrollment
  Evaluate the intensity of 99mTc-MIP-1404 uptake with respect to PSMA expression

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Slawin, M.D., Principal Investigator — Vanguard Urologic Research Foundation, University of Texas, Houston
Locations (1):
- The University of Texas Health Science Center - Houston, Houston, Texas, United States

REFERENCES:
- [Background] Pinto JT, Suffoletto BP, Berzin TM, Qiao CH, Lin S, Tong WP, May F, Mukherjee B, Heston WD. Prostate-specific membrane antigen: a novel folate hydrolase in human prostatic carcinoma cells. Clin Cancer Res. 1996 Sep;2(9):1445-51. PMID 9816319
- [Background] Smith-Jones PM, Vallabahajosula S, Goldsmith SJ, Navarro V, Hunter CJ, Bastidas D, Bander NH. In vitro characterization of radiolabeled monoclonal antibodies specific for the extracellular domain of prostate-specific membrane antigen. Cancer Res. 2000 Sep 15;60(18):5237-43. PMID 11016653
- [Background] Ghosh A, Heston WD. Tumor target prostate specific membrane antigen (PSMA) and its regulation in prostate cancer. J Cell Biochem. 2004 Feb 15;91(3):528-39. doi: 10.1002/jcb.10661. PMID 14755683
- [Background] Kinoshita Y, Kuratsukuri K, Landas S, Imaida K, Rovito PM Jr, Wang CY, Haas GP. Expression of prostate-specific membrane antigen in normal and malignant human tissues. World J Surg. 2006 Apr;30(4):628-36. doi: 10.1007/s00268-005-0544-5. PMID 16555021
- [Background] Murphy GP, Elgamal AA, Su SL, Bostwick DG, Holmes EH. Current evaluation of the tissue localization and diagnostic utility of prostate specific membrane antigen. Cancer. 1998 Dec 1;83(11):2259-69. PMID 9840525
- [Background] Milowsky MI, Nanus DM, Kostakoglu L, Sheehan CE, Vallabhajosula S, Goldsmith SJ, Ross JS, Bander NH. Vascular targeted therapy with anti-prostate-specific membrane antigen monoclonal antibody J591 in advanced solid tumors. J Clin Oncol. 2007 Feb 10;25(5):540-7. doi: 10.1200/JCO.2006.07.8097. PMID 17290063
- [Background] Vallabhajosula S, Kuji I, Hamacher KA, Konishi S, Kostakoglu L, Kothari PA, Milowski MI, Nanus DM, Bander NH, Goldsmith SJ. Pharmacokinetics and biodistribution of 111In- and 177Lu-labeled J591 antibody specific for prostate-specific membrane antigen: prediction of 90Y-J591 radiation dosimetry based on 111In or 177Lu? J Nucl Med. 2005 Apr;46(4):634-41. PMID 15809486
- [Background] Hillier SM, Maresca KP, Femia FJ, Marquis JC, Foss CA, Nguyen N, Zimmerman CN, Barrett JA, Eckelman WC, Pomper MG, Joyal JL, Babich JW. Preclinical evaluation of novel glutamate-urea-lysine analogues that target prostate-specific membrane antigen as molecular imaging pharmaceuticals for prostate cancer. Cancer Res. 2009 Sep 1;69(17):6932-40. doi: 10.1158/0008-5472.CAN-09-1682. Epub 2009 Aug 25. PMID 19706750
- [Background] Olson WC, Heston WD, Rajasekaran AK. Clinical trials of cancer therapies targeting prostate-specific membrane antigen. Rev Recent Clin Trials. 2007 Sep;2(3):182-90. doi: 10.2174/157488707781662724. PMID 18474004
- [Background] Rajasekaran AK, Anilkumar G, Christiansen JJ. Is prostate-specific membrane antigen a multifunctional protein? Am J Physiol Cell Physiol. 2005 May;288(5):C975-81. doi: 10.1152/ajpcell.00506.2004. PMID 15840561
- [Background] Slovin SF. Targeting novel antigens for prostate cancer treatment: focus on prostate-specific membrane antigen. Expert Opin Ther Targets. 2005 Jun;9(3):561-70. doi: 10.1517/14728222.9.3.561. PMID 15948673
- [Background] Wang X, Yin L, Rao P, Stein R, Harsch KM, Lee Z, Heston WD. Targeted treatment of prostate cancer. J Cell Biochem. 2007 Oct 15;102(3):571-9. doi: 10.1002/jcb.21491. PMID 17685433
- [Background] Barrett PH, Bell BM, Cobelli C, Golde H, Schumitzky A, Vicini P, Foster DM. SAAM II: Simulation, Analysis, and Modeling Software for tracer and pharmacokinetic studies. Metabolism. 1998 Apr;47(4):484-92. doi: 10.1016/s0026-0495(98)90064-6. PMID 9550550
- [Background] Stabin MG, Siegel JA. Physical models and dose factors for use in internal dose assessment. Health Phys. 2003 Sep;85(3):294-310. doi: 10.1097/00004032-200309000-00006. PMID 12938720
- [Background] Stabin MG, Sparks RB, Crowe E. OLINDA/EXM: the second-generation personal computer software for internal dose assessment in nuclear medicine. J Nucl Med. 2005 Jun;46(6):1023-7. PMID 15937315
- [Background] Pan ZY, Wolf W. Computer package for the calculation of the radiation dose to patients, based on the MIRD approach. J Nucl Med. 1985 Mar;26(3):318-20. No abstract available. PMID 3882906